CLINICAL TRIAL: NCT06970899
Title: Evaluation of the CycloPE® Device Used in Patients With a Suspected Bloodstream Infection
Brief Title: Initial Feasibility Study of the CycloPE® Device
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PATH EX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QMS-CIP-101
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Infection; Bacteremia Sepsis; Systemic Inflammatory Response Syndrome (SIRS)
MeSH Terms: conditions — Sepsis; Infections; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- PATH EX CycloPE® Device (Experimental): Treated with PATH EX CycloPE® Device
  Interventions: Device: PATH EX CycloPE® Device

INTERVENTIONS:
Device: PATH EX CycloPE® Device — Participants in this arm will receive two extracorporeal blood filtration treatments using the PATH EX CycloPE® device. The first treatment will be initiated following baseline assessments, and the second treatment will occur 24-36 hours after the start of the first treatment. Each treatment will last up to 4 hours. The device is designed to target and remove bacteria from the bloodstream. All participants will also receive standard-of-care treatment for sepsis, including IV antibiotics, as determined by the treating physician.

SUMMARY:
This is a single-center, prospective, single-arm clinical study to evaluate the feasibility, safety, and performance of the PATH EX CycloPE® device on suspected bacteremia-associated sepsis. All participants are adults diagnosed with suspected bacteremia-associated sepsis, admitted to the intensive care unit (ICU), and meet the inclusion criteria.

DETAILED DESCRIPTION:
This is a single-center, prospective, single-arm clinical study designed to evaluate the feasibility, safety, and performance of the PATH EX CycloPE® device for the treatment of suspected bacteremia-associated sepsis in critically ill patients. Participants in the study will be adults diagnosed with suspected bacteremia-associated sepsis, admitted to the intensive care unit (ICU), and meeting all inclusion and exclusion criteria. Each patient will undergo two treatments with the PATH EX CycloPE® device. The second treatment will occur 24-36 hours after the start of the first treatment, with each session lasting 4 hours. Clinical and laboratory assessments will be conducted at baseline and predefined intervals during and after the treatment period to monitor safety and evaluate the device's performance.

The primary endpoints focus on feasibility and safety, including device-related adverse events and procedural success. Secondary endpoints will assess infection resolution through microbial eradication, reductions in biomarkers, and changes in hematology and chemistry indices.

The PATH EX CycloPE® device is a novel extracorporeal blood filtration system designed to directly target and remove bacteria from the bloodstream. By addressing the root cause of sepsis, the device has the potential to improve outcomes for critically ill patients.

This study will generate critical data to inform the design of future clinical trials and support the development of this breakthrough technology for the treatment of sepsis. All data will be collected, analyzed, and reported in compliance with Good Clinical Practice (GCP) guidelines and applicable regulatory requirements

ELIGIBILITY:
Inclusion Criteria: 1. Hospitalized adults (age >= 18 years, male and female) 2. Receiving IV antibiotic therapy 3. Presence of at least 2 of the 4 SIRS criteria:

1. Body temperature > 101°F (38.3°C) or < 96.8°F (36°C);
2. Heart rate > 90 beats per minute;
3. Respiratory rate > 20 breaths per minute;
4. White blood cell count > 12,000/mm³, < 4,000/mm³, or > 10% bands 4. Clinical evidence of new organ dysfunction 5. Procalcitonin (PCT) levels ≥ 0.5 ng/mL

Exclusion Criteria: 1. Inability to maintain a minimum mean arterial pressure of ≥ 65 mmHg despite vasopressor therapy and fluid resuscitation 2. Medical conditions requiring regular blood transfusion 3. Active bleeding (e.g., active GI bleeding, hematuria or epistaxis, untreated coagulopathy or bleeding from a non-compressible site) 4. Absolute neutrophil count less than 500 cells/mm3 5. Platelet count less than 50,000 cells/mm3 6. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period 7. Known hypersensitivity to Polymyxin E 8. Known hypersensitivity to Vancomycin 9. Subject has known sensitivity/allergy to heparin or has a history of heparin induced thrombocytopenia (HIT) 10. IV antibiotic treatment initiated > 48 hours before baseline screening

This exclusion criterion is not applicable for two cases:

1. IV antibiotic treatment initiated > 48 hours before baseline screening has been deemed ineffective based on the clinical judgment of the investigator.
2. If the patient has discontinued IV antibiotic therapy for a continuous period of 24 hours or more within the 48-hour window immediately preceding baseline screening.

   11. Participated in an interventional clinical study within 28 days prior to Day 0 or undergoing treatment anticipated to require significant blood draws 12. Have been previously enrolled in this clinical trial 13. History of or known hypercoagulable state 14. Known history of a condition that may result in an increased risk for thrombosis 15. Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate for enrollment 16. Unable to obtain informed consent from either patient or legally authorized representative 17. Patients who cannot tolerate placement of double-lumen catheter 18. Suspected or confirmed SARS-CoV-2 infection (COVID-19) that cannot be resolved before administration of investigational device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events (SAEs) related to the investigational device | 7 days
  The incidence and nature of serious adverse events (SAEs) that are related to the use of the PATH EX CycloPE® device will be assessed to evaluate the safety of the investigational device.

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs) not related to the investigational device or procedure | 7 days
  The incidence of SAEs occurring while connected to the device that are not deemed related to the investigational device or procedure will be assessed.
Clinically significant changes in hematology indices | 7 days
  Clinically significant changes in hematology indices will be evaluated to monitor potential safety concerns.
Clinically significant changes in chemistry indices | 7 days
  Clinically significant changes in chemistry indices will be evaluated to monitor potential safety concerns.
Device deficiencies and malfunctions | 7 days
  Any deficiencies or malfunctions of the PATH EX CycloPE® device, including procedural or technical issues, will be recorded and analyzed.
Clinical and laboratory adverse events (AEs) | 7 days
  The incidence of all clinical and laboratory adverse events (AEs) occurring up to 7 days post-enrollment will be assessed for potential safety concerns.
Pathogen reduction in the bloodstream | 7 days
  Pathogen reduction will be evaluated by measuring the increase in time to positivity (TTP) of blood samples before versus after treatment with the PATH EX CycloPE® device. Only blood samples with a measurable positive TTP before treatment will be included in this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Harutyun N Mangoyan, MD. PhD, Principal Investigator — Erebuni Medical Center
Locations (1):
- Erebuni Medical Cener, Yerevan, Armenia, Armenia

IPD SHARING:
Plan to Share IPD: No